CLINICAL TRIAL: NCT04547387
Title: Carotid Artery Revascularization Using TransCarotid flOw Reversal Cerebral Protection And CGUARD MicroNET-Covered Embolic Prevention Stent System to Reduce Strokes in Patients With Symptoms or Signs of Cerebral Ischemia: TOP-GUARD Study
Brief Title: TCAR Cerebral Protection And MicroNET-Covered Stent To Reduce Strokes
Acronym: TOP-GUARD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John Paul II Hospital, Krakow (Other)
Responsible Party: Sponsor
Other Study IDs: TOP-GUARD
Record Dates: First submitted 2020-08-31; First posted 2020-09-14 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid Artery Stenting: Consecutive patients with symptoms or signs of ischemic cerebral injury eligible for endovascular carotid artery revascularization using direct carotid artery access and MicroNET covered carotid stent plaque exclusion under cerebral protection by temporary flow reversal
  Interventions: Device: Trans-carotid access revascularization with MicroNET covered stent implantation

INTERVENTIONS:
Device: Trans-carotid access revascularization with MicroNET covered stent implantation — Implantation of the micronet covered self-expanding carotid stent during temporary cerebral flow reversal achieved with direct common carotid artery puncture

SUMMARY:
Prospective, single center clinical study in consecutive patients with symptoms or signs of carotid stenosis related ischemic cerebral injury undergoing carotid revascularization in primary and secondary stroke prevention. MicroNET-covered stent is implanted using direct carotid artery access and temporary flow reversal to combine optimal intraprocedural cerebral protection and optimal plaque exclusion.

DETAILED DESCRIPTION:
Prospective, single-center clinical study in consecutive patients undergoing carotid revascularization with MicroNET-covered stent implanted through direct carotid artery access with temporary, intraprocedural flow reversal neuroprotection to provide primary and secondary stroke prevention.

It is an open-label, non-randomized single-arm study supported by the grant from Jagiellonian University Medical college (K/ZDS/007819).

Stroke is a major health problem affecting individual patients and their families and entire societies with death and disability impact (fundamental disability cause in Poland, Europe, and the USA). Atherosclerotic carotid artery stenosis plays an important part in a stroke etiology through embolic and/or hemodynamic mechanism).

Endovascular treatment with first-generation carotid stents is inherently related to plaque and thrombus prolapse through stent struts, as confirmed with the intravascular imaging (IVUS and OCT), and monitoring of cerebral embolism by DW-MRI. Plaque prolapse related embolism may occur after neuroprotection device removal. Postprocedural plaque-prolapse related ischemic events are responsible for 40-60% complications up to 30 days, as indicated by 30-day results of large clinical trials (CAPTURE, CREST, or ICSS).

A successful attempt to address this problem has been an introduction and routine use of MicroNET-covered stent. The MicroNET attached to the metallic stent prevents intraluminal plaque prolapse. MRI imaging indicated a significant reduction of intraprocedural embolism and near-elimination of post-procedural brain embolism by CGuard application. Clinical research and meta-analysis of studies confirmed the safety and efficacy of the stent. Consistent results were demonstrated in registries such as PARADIGM.

Another critical approach in increasing the safety of the endovascular route of carotid revascularization is development and increased clinical uptake of minimally invasive endovascular strategies is the direct common carotid artery access for stenting procedures. This way, one can avoid femoral cannulation and navigation through the aorta and aortic arch branches. Trans-Carotid Arterial Revascularization (TCAR) offers a neuroprotection mechanism by a temporary reversal of the cerebral flow similar to Mo.Ma Ultra or GORE Flow Reversal systems, but without limitations of femoral access and aortic arch cannulation. TCAR system was CE marked in 2014, and more than 20 000 TCAR procedures were performed worldwide. A recent analysis by Yee et al. demonstrated that TCAR carotid stenting procedures are equivalent to surgical endarterectomy regarding safety and efficacy, but with lower invasiveness, avoiding the aortic arch (and its cannulation-related cerebral embolism) and shortened procedure time.

According to published studies and our own experience, proximal neuroprotection, and in particular, the one achieved through direct carotid artery access, minimizes cerebral (micro)embolization risk.

Our prospective TOP-GUARD study aims to evaluate early-, mid- and longterm outcome data (up to 5 years) on the results of carotid revascularization combining two systems that are currently considered safest: temporary cerebral flow-reversal during stent introduction via direct carotid artery access and MicroNET-covered stent implantation.

Both systems are CE-marked (from 2014), have been successfully used in our center, and will follow their on-label indications.

The TCAR system from SilkRoad Medical (EnRoute) is the preferred method to obtain flow reversal for transcervical CAS in the study. However, due to interruption of the EnRoute system supplies (COVID19, SARS-CoV-2 Pandemic), routinely available sheaths, catheters, and blood filters may be used according to literature to assemble the flow reversal circuit, enabling continuation of the study as per the Ethical Committee updated approval.

Consecutive patients with symptoms or signs of cerebral ischemia (ie. patients with an increased risk of complications when conventional carotid stents and neuroprotection systems are used) will undergo NeuroVascular Team (neurologist, interventionalist, and vascular surgeon) evaluation for their eligibility. They will be treated according to the center standard of care, including necessary peri- and postprocedural medication.

MRI cerebral imaging will be performed at baseline, 24-48 hours post-procedurally and at 90 days in 50% of study participants.

ELIGIBILITY:
General Inclusion Criteria:

* Consecutive adult patients with clinical symptoms and/or signs (on cerebral imaging) of of carotid stenosis-related cerebral ischemic injury eligible for TCAR carotid revascularization according to NeuroVascular Team evaluation and local standards
* Symptomatic and asymptomatic carotid artery stenosis with ipsilateral ischemic lesions in brain imaging (CT or MRI)
* Informed written consent
* Declared compliance and consent to adhere to scheduled follow up and routine long term follow up

Angiographic Inclusion Criteria:

* De novo or neo-atherosclerotic carotid artery lesion
* NASCET criteria ≥50% carotid artery stenosis in patients with ipsilateral TIA, stroke or amaurosis fugax within last 6 months
* NASCET criteria ≥70-80% carotid artery stenosis in asymptomatic patients especially with ipsilateral ischemic lesions in brain imaging (CT or MRI)

General Exclusion Criteria:

* Lack of technical feasibility or logistic opportunity to perform procedure (device availability)
* Life expectancy less than 1 year
* Renal insufficiency with creatinine >3mg/dL
* Myocardial infarction within last 72 hours before procedure
* Pregnant women
* Coagulopathies
* Allergy to contrast media not amenable to pharmacotherapy

Angiographic Exclusion Criteria:

* Total carotid artery occlusion
* Stent in the carotid artery preventing artery cannulation or introduction of stent or protective device
* Anatomic variants preventing introduction of stent or protective device
* Significant common carotid artery stenosis proximal to target vessel
* Moving plaque in aortic arch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comer study in consecutive increased-risk patients (defined as those with symptoms or signs of carotid stenosis-related cerebral ischemic injury) eligible for trans-carotid access proximal cerebral protection and MicroNET-covered stent implantation based on the NeuroVascular Team evaluation and agreemment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Immediate procedural success rate | 48 hours or hospital discharge, whatever comes first
  Combined endpoint of TECHNICAL SUCCESS (insertion and removal of the embolic protection device, successful stent delivery, implantation and delivery system retrieval, with residual stenosis ≤30%) AND CLINICAL SUCCESS (freedom from MACNE (death, stroke, myocardial infarction) up to 48 hrs or hospital discharge)

SECONDARY OUTCOMES:
Freedom from MACNE up to 30 days | 30 days postprocedural
  Freedom from MACNE (death, ipsi- and contralateral stroke, myocardial infarction)
Freedom from MACNE up to 90 days | 90 days postprocedural
  Freedom from MACNE (death, ipsi- and contralateral stroke, myocardial infarction)
Occurence of new, postprocedural ipsilateral DW-MRI ischemic lesions | 48 hours post procedure
  Occurence of new, postprocedural ipsilateral DW-MRI ischemic lesions (evaluated in 50% of eligible study population)
Occurence of new, postprocedural ipsilateral DW-MRI ischemic lesions | 90 days post procedure
  Occurence of new, postprocedural ipsilateral DW-MRI ischemic lesions (non-contrast evaluation in 50% of eligible study population)
Rate of complete stent expansion and apposition | During procedure
  Complete stent expansion and apposition on IVUS (if performed) in absence of plaque prolapse
Rate of ipsilateral stroke | 30 days to 1 year post procedure
  Rate of ipsilateral stroke
Rate of ipsilateral stroke | 1 year to 5 years post procedure
  Rate of ipsilateral stroke
Rate of any stroke | Up to 5 years post procedure
  Rate of any stroke
Stroke free survival | Up to 5 years post procedure
  Stroke free survival
Ipsilateral stroke free survival | Up to 5 years post procedure
  Ipsilateral stroke free survival
Rate of target vessel restenosis requiring treatment | Up to 5 years post procedure
  Rate of target vessel restenosis requiring treatment
Ultrasound measured Peak Systolic Velocity in target artery | 48 hours post procedure
  Ultrasound measured Peak Systolic Velocity in target artery
Ultrasound measured Peak Systolic Velocity in target artery | At 30 days post-procedure
  Ultrasound measured Peak Systolic Velocity in target artery
Ultrasound measured Peak Systolic Velocity in target artery | At 1 year post-procedure
  Ultrasound measured Peak Systolic Velocity in target artery

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, DPhil, Principal Investigator — Department of Cardiac and Vascular Diseases, John Paul II Hospital; Mariusz Trystula, MD, PhD, Principal Investigator — Department of Vascular Surgery, John Paul II Hospital
Locations (1):
- Department of Cardiac and Vascular Diseases, John Paul II Hospital, Krakow, Maloplska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yee EJ, Wang SK, Timsina LR, Ruiz-Herrera S, Liao JL, Donde NN, Fajardo AC, Motaganahalli RL. Propensity-Matched Outcomes of Transcarotid Artery Revascularization Versus Carotid Endarterectomy. J Surg Res. 2020 Aug;252:22-29. doi: 10.1016/j.jss.2019.12.003. Epub 2020 Mar 26. PMID 32222590
- [Background] Musialek P, Mazurek A, Trystula M, Borratynska A, Lesniak-Sobelga A, Urbanczyk M, Banys RP, Brzychczy A, Zajdel W, Partyka L, Zmudka K, Podolec P. Novel PARADIGM in carotid revascularisation: Prospective evaluation of All-comer peRcutaneous cArotiD revascularisation in symptomatic and Increased-risk asymptomatic carotid artery stenosis using CGuard MicroNet-covered embolic prevention stent system. EuroIntervention. 2016 Aug 5;12(5):e658-70. doi: 10.4244/EIJY16M05_02. PMID 27180302
- [Background] Mazurek A, Borratynska A, Malinowski KP, Brozda M, Gancarczyk U, Dluzniewska N, Czyz L, Duplicka M, Sobieraj E, Trystula M, Drazkiewicz T, Podolec P, Musialek P. MicroNET-covered stents for embolic prevention in patients undergoing carotid revascularisation: twelve-month outcomes from the PARADIGM study. EuroIntervention. 2020 Dec 4;16(11):e950-e952. doi: 10.4244/EIJ-D-19-01014. No abstract available. PMID 32482614
- [Background] Chang DW, Schubart PJ, Veith FJ, Zarins CK. A new approach to carotid angioplasty and stenting with transcervical occlusion and protective shunting: Why it may be a better carotid artery intervention. J Vasc Surg. 2004 May;39(5):994-1002. doi: 10.1016/j.jvs.2004.01.045. PMID 15111851
- [Background] Criado E, Fontcuberta J, Orgaz A, Flores A, Doblas M. Transcervical carotid stenting with carotid artery flow reversal: 3-year follow-up of 103 stents. J Vasc Surg. 2007 Nov;46(5):864-9. doi: 10.1016/j.jvs.2007.07.028. PMID 17980271
- [Background] Pipinos II, Johanning JM, Pham CN, Soundararajan K, Lynch TG. Transcervical approach with protective flow reversal for carotid angioplasty and stenting. J Endovasc Ther. 2005 Aug;12(4):446-53. doi: 10.1583/05-1561.1. PMID 16048376
- [Derived] Trystula M, VAN Herzeele I, Kolvenbach R, Tekieli L, Fonteyne C, Mazurek A, Dzierwa K, Chmiel J, Lindsay J, Kwiatkowski T, Hydzik A, Oplawski M, Bederski K, Musialek P. Next-generation transcarotid artery revascularization: TransCarotid flOw Reversal Cerebral Protection And CGUARD MicroNET-Covered Embolic Prevention Stent System To Reduce Strokes - TOPGUARD Study. J Cardiovasc Surg (Torino). 2024 Jun;65(3):181-194. doi: 10.23736/S0021-9509.24.13121-7. PMID 39007552